CLINICAL TRIAL: NCT05691764
Title: Effect of Cyclosporine and Remote Ischemic Preconditioning on MDA, Calcium Cytosol Concentration, and Mitochondrial Edema in Reperfusion Ischemia Injury: Research on Tetralogy Fallot Patients With Correction Surgery
Brief Title: Effect of Cyclosporine and Remote Ischemic Preconditioning in Reperfusion Ischemia Injury on Tetralogy Fallot Patients With Correction Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Jefferson K Hidayat, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IndonesiaUAnes055
Record Dates: First submitted 2022-12-15; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Myocardial Injury; Cardiac Surgery
Keywords: RIPC; cyclosporine; ischemia reperfusion injury; MDA; calcium cytosol; tetralogy Fallot; mitochondrial edema; infundibulum
MeSH Terms: conditions — Reperfusion Injury; Tetralogy of Fallot | interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyclosporin + RIPC (Experimental): This group received cyclosporin intravenously 2 hours pre-induction of anesthesia, with the dose of 3 mg/ kg body weight. RIPC was performed preoperatively after induction of anesthesia by inflating pressure cuff on the extremity 30 mmHg higher than systolic blood pressure of the patient for 5x5 minutes with 5 minutes reperfusion interval.
  Interventions: Drug: Cyclosporin; Procedure: remote ischemic preconditioning
- Control (Placebo Comparator): This group received placebo intravenously 2 hours pre-induction of anesthesia.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cyclosporin — Cyclosporin was administered intravenously with the dose of 3 mg/ kg body weight
  Other Names: Sandimmun
  Arms: Cyclosporin + RIPC
Procedure: remote ischemic preconditioning — Performed by inflating pressure cuff on the extremity 30 mmHg higher than systolic blood pressure of the patient for 5x5 minutes with 5 minutes reperfusion interval
  Other Names: RIPC
  Arms: Cyclosporin + RIPC
Drug: Placebo — Intravenous placebo
  Arms: Control

SUMMARY:
The study aimed to evaluate the combined effects of cyclosporine and remote ischemic preconditioning on MDA, calcium cytosol concentration, and mitochondrial edema in tetralogy Fallot patients undergoing corrective surgery.

DETAILED DESCRIPTION:
Forty patients undergoing tetralogy Fallot corrective surgery were randomized to RIPC and cyclosporine (n=20) and control (n=20). Cyclosporin was administered 2 hour pre induction of anesthesia with the dose of 3 mg/kg body weight intravenously. RIPC was performed preoperatively after induction of anesthesia by inflating pressure cuff on the extremity 30 mmHg higher than systolic blood pressure of the patient for 5x5 minutes with 5 minutes reperfusion interval. Blood samples from coronary sinus and biopsies from the myocardial infundibulum were obtained three times at the condition of pre ischemic, ischemic, and reperfusion. MDA was measured from the blood samples, meanwhile calcium cytosol concentration and mitochondrial edema was measured from the biopsy samples.

ELIGIBILITY:
Inclusion Criteria:

* Tetralogy Fallot patient that is undergoing correction surgery
* Has an ideal anatomy for corrective surgery, namely: Pulmonary artery size within normal limits (according to the kirklin table), Mc Goon ratio> 1.5, Nakata index> 200, normal coronary artery ostium and good biventricular function.

Exclusion Criteria:

* Patient refuses the procedure
* Patient with acute kidney injury
* Patient without lower extremity
* Patient with cyclosporin allergy

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Malondialdehyde (MDA) | 1 year
  ROS level is determined by measuring MDA concentration (nmol/mL)
Calcium cytosol concentration | 1 year
  Calcium concentration (nmol/mL) in cytosol is determined by ratiometric analysis on Fura Red- dyed heart cells.
Mitochondrial edema | 1 year
  Mitochondrial edema (%) is measured by decreasing of optical density that indicates change in mitochondrial matrix volume.

SECONDARY OUTCOMES:
Cardiac index | 1 year
  Examined with echocardiography, unit of measurement is litres per minute per square metre (L/min/m2).
Troponin I | 1 year
  Measured from venous blood, unit of measurement is nanograms per milliliter (ng/mL).
Creatine kinase- MB (CKMB) | 1 year
  Measured from venous blood, unit of measurement is units per liter (IU/L).
Vasoactive inotropic score (VIS) | 1 year
  VIS was calculated as: dopamine dose (μg/kg/min) + dobutamine dose (μg/kg/min) + 100 × epinephrine dose (μg/kg/min) + 10 × milrinone dose (μg/kg/min) + 10 000 × vasopressin dose (unit/kg/min) + 100 × norepinephrine dose (μg/kg/min).

CONTACTS AND LOCATIONS:
Overall Officials: Jefferson K Hidayat, MD, Principal Investigator — Indonesia University
Locations (1):
- Indonesia University, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu Q, Wang T, Chen S, Zhou Q, Li H, Hu N, Feng Y, Dong N, Yao S, Xia Z. Cardiac protective effects of remote ischaemic preconditioning in children undergoing tetralogy of fallot repair surgery: a randomized controlled trial. Eur Heart J. 2018 Mar 21;39(12):1028-1037. doi: 10.1093/eurheartj/ehx030. PMID 28329231
- [Result] Davidson SM, Ferdinandy P, Andreadou I, Botker HE, Heusch G, Ibanez B, Ovize M, Schulz R, Yellon DM, Hausenloy DJ, Garcia-Dorado D; CARDIOPROTECTION COST Action (CA16225). Multitarget Strategies to Reduce Myocardial Ischemia/Reperfusion Injury: JACC Review Topic of the Week. J Am Coll Cardiol. 2019 Jan 8;73(1):89-99. doi: 10.1016/j.jacc.2018.09.086. PMID 30621955
- [Result] Zalewski J, Claus P, Bogaert J, Driessche NV, Driesen RB, Galan DT, Sipido KR, Buszman P, Milewski K, Van de Werf F. Cyclosporine A reduces microvascular obstruction and preserves left ventricular function deterioration following myocardial ischemia and reperfusion. Basic Res Cardiol. 2015 Mar;110(2):18. doi: 10.1007/s00395-015-0475-8. Epub 2015 Feb 27. PMID 25720581
- [Result] Chen HW, Chien CT, Yu SL, Lee YT, Chen WJ. Cyclosporine A regulate oxidative stress-induced apoptosis in cardiomyocytes: mechanisms via ROS generation, iNOS and Hsp70. Br J Pharmacol. 2002 Nov;137(6):771-81. doi: 10.1038/sj.bjp.0704908. PMID 12411407